CLINICAL TRIAL: NCT04415372
Title: Macromolecular Imaging of White and Gray Matter Pathology in Multiple Sclerosis
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0310; 1R01EB027087-01 (NIH); A539300 (Other: University of Wisconsin, Madison); SMPH/RADIOLOGY/RADIOLOGY (Other: University of Wisconsin, Madison); Protocol Version 4/8/2024 (Other: UW Madison)
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis; MS
Keywords: Magnetic resonance imaging
MeSH Terms: conditions — Multiple Sclerosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Cognitive Impairment: Adults diagnosed with MS that have evidence of cognitive decline.
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Neuropsychological Testing
- No Cognitive Impairment: Adults diagnosed with MS that have no evidence of cognitive decline.
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Neuropsychological Testing
- Healthy Controls: Healthy adult volunteers will form a control group matched for age, gender, education, handedness
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — The MRI protocol will include conventional testing for MS lesion detection and functional MR imaging to localize associated neurocognitive domains in each subject.
  Other Names: Functional MRI
Diagnostic Test: Neuropsychological Testing — A comprehensive battery of neuropsychological tests will be administered to assess memory, new learning, spatial processing and higher executive function.
  Groups: Cognitive Impairment; No Cognitive Impairment

SUMMARY:
The overall purpose of this research is to determine whether new macromolecular measures optimized for whole brain (gray matter and white matter) magnetic resonance imaging (MRI), predict neuro-cognitive impairment in multiple sclerosis (MS) patients.

DETAILED DESCRIPTION:
MRI is a vital component of a MS work-up, providing noninvasive evidence of MS lesions, detecting active inflammatory lesions, and measuring brain atrophy to assess neurodegeneration. Recent years of MRI research have generated strong evidence of gray matter (GM) involvement in MS, resulting in the reclassification of MS as a whole-brain disease. Similar to white matter (WM), a primary target of MS pathology in GM is myelin, the protective sheath insulating the penetrating axons within GM and extending brain connectivity all the way to the neuronal bodies.

This aim of this research is to examine if the associations between imaging measures of GM disease and cognitive performance can establish GM-based imaging correlates predicting the disease course and accurately assessing treatment results.

This observational research will enroll adults diagnosed with MS both with and without cognitive impairment. Subjects will be asked to complete a single research visit that includes the administration of a MRI scan and a neuro-cognitive testing session.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite MS
* Adult age 18 to 60

Exclusion Criteria:

* Contraindication to MRI
* Changes in MS therapy in the last 6 months
* Less than 6 weeks after relapse or corticosteroid use
* Currently taking medication that may affect cognition (e.g. donepezil, rivastigmine, adderall)
* History of significant alcohol or drug abuse
* Current or recent significant migraines
* Confounding neurological or cognitive disorders or deficits (stroke, Parkinson's disease, Alzheimer's disease, epilepsy)
* Sensory or physical impairments that might interfere significantly with cognitive testing
* History of developmental or learning disability or attention-deficit/hyperactivity disorder.\

Exclusion Criteria for Healthy Controls:

* history of alcohol/drug abuse
* history of migraines
* developmental or learning disability/attention-deficit/hyperactivity disorder
* currently pregnant/breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults diagnosed with MS both with and without evidence of cognitive impairment.
  Healthy controls will be recruited from the MRI Volunteer Database (2017-0004, PI: Reeder)
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Measurement of macromolecular proton content (MPC) by Magnetic resonance imaging | 24 hours
  Macromolecular Proton Fraction (MPF) is calculated from several specially acquired MR images and is characterized by high degree of sensitivity and specificity to tissue macromolecules, which are the main target of pathological process in neurodegenerative diseases including multiple sclerosis (MS). These properties of MPF are in contrast with standard MR images, which are primarily sensitive to tissue water molecules.

SECONDARY OUTCOMES:
Neurocognitive performance as measured by Minimal Assessment of Cognitive Function in MS (MACFIMS) battery of neuropsychological (NP) tests | 24 hours
  The results of Minimal Assessment of Cognitive Function in MS (MACFIMS) battery of neuropsychological (NP) tests will form the secondary outcome measure. The NP scores will be correlated with MPF to study association between macromolecular tissue damage and neurocognitive performance.
Neurocognitive performance as measured by the Montreal Cognitive Assessment (MoCA) score | 24 hours
  Neurocognitive performance will be measured by Montreal Cognitive Assessment. MoCA scores range from 0 to 30, higher values corresponding to better cognitive performances.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Samsonov, PhD, Principal Investigator — UW Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No